CLINICAL TRIAL: NCT05480696
Title: The Efficacy of Soluble Fibre Supplementation for the Treatment of Pediatric Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Soluble Fibre Supplementation in NAFLD
Acronym: FIND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14888; 471270 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2022-07-22; First posted 2022-07-29 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis; Hepatic Steatosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly allocated (1:1) to the OF+INU supplementation (intervention) or placebo group in a concealed fashion using REDCap databases, generated by a computer algorithm in permuted blocks of 2 and 4, to avoid imbalances. Study investigators and participants will be blinded to group allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oligofructose Inulin Supplementation (Experimental): The intervention group will receive a daily fibre supplementation of (fructo-oligosaccharide enriched inulin, 4g twice daily; Orafti®Synergy1, BENEO), a tasteless white powder contained within a tear-able, partitioned 4g sachet, sprinkled and dissolved in 125 mL of water.
  Interventions: Dietary Supplement: Fructo-oligosaccharide enriched inulin supplement
- Maltodextrin Supplementation (Sham Comparator): The control group will receive a daily supplementation of carbohydrate placebo (isocaloric maltodextrin), identical in colour, packaging, preparation, and dose (4g, twice daily; C*Dry MD™,Cargill).
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Fructo-oligosaccharide enriched inulin supplement — Experiment
  Arms: Oligofructose Inulin Supplementation
Other: Maltodextrin — Placebo.
  Arms: Maltodextrin Supplementation

SUMMARY:
The FIND study will look at the effect of a nutritional mixed fibre supplement, oligofructose and inulin (OF+INU), on children with non-alcoholic fatty liver disease. In this randomized, double- blind controlled trial, subjects will be given a supplement, in the form of oral pills, and will have bloodwork performed, their diets analyzed, and liver fat measured at several timepoints. Liver fat will be measured by using a specialized MRI device located at St. Joseph's Hospital. Subjects will be recruited from the Children's Exercise and Nutrition Clinic.

DETAILED DESCRIPTION:
The FIND (Fibre in Non-Alcoholic Fatty Liver Disease) study will be a single-centre, randomized, double-blind placebo-controlled trial comparing the effects of 6 months of mixed oligofructose and inulin (OF+INU) supplementation vs placebo on hepatic fat content, hepatic stiffness, metabolic outcomes, and body composition in children ages 8-17 years old.

Assessments such as MRI measurements of hepatic fat and hepatic stiffness, anthropometry and pubertal status questionnaires, and other investigations such as body composition via dual energy X-ray absorptiometry (DXA), fasting lipids, liver enzymes, blood glucose and oral-glucose tolerance (OGTT) tests will be performed; and randomization will be conducted via REDCap software.

Eighty participants will be enrolled for baseline evaluation in order to randomize sixty participants for the intervention phase (i.e. thirty participants per study group). Participants will consume one packet (4g) of OF+INU or placebo (Maltodextrin) daily. If tolerated, this will increase to one packet twice daily. Several strategies will be implemented to increase compliance, including text message reminders (daily for first week, then weekly), study calls to assess compliance and tolerability, and check-ins with participants at each clinic visit. These interactions will allow the study team to assess challenges and offer prompt support. Compliance will be assessed at each study visit by counting empty and unused sachets. Treatment with OF+INU or placebo will occur for 6 months, with study visits being conducted at baseline evaluation, 3 months and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-17 years
* Diagnosed with obesity (BMI ≥2 standard deviations above WHO reference median)
* Enrolled in GHWM Clinic
* Clinical evidence of NAFLD (elevation of ALT, greater than 2x upper-limit-of-normal (ULN) [ALT>80 IU/L for 8-17 years of age], and hepatic steatosis measured as part of clinic enrolment).

Exclusion Criteria:

* Type 1, Type 2 diabetes mellitus (T1DM, T2DM)
* Contraindications to having MRI (claustrophobia, metal implant, recent tattoo, weight > 300lbs)
* Concomitant use of other fibre supplements
* Medications known to affect hepatic fat content, taken within the past year (i.e., glucocorticoids, anabolic steroids, tetracycline, anticonvulsants, antipsychotics, glucose- lowering medications)
* Presence of another known cause of liver disease
* Known allergy or hypersensitivity to OF-INU supplementation
* Self-reported alcohol intake >7 drinks/week or 3 drinks/day

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in hepatic fat content. | Six months
  Hepatic fat content will be measured via MRI at baseline and 6-months using standard techniques, optimized for accuracy, precision and reproducibility of proton density fat fraction (PDFF) quantification.

SECONDARY OUTCOMES:
Change in hepatic stiffness. | Six months
  Hepatic stiffness, a measure of hepatic fibrosis, will be measured via MRI using standard techniques.
Change in glycemic control, or insulin resistance. | Six months
  Measured using plasma glucose (fasting and + 2 hours following oral glucose load) and HbA1c from a 2-hour OGTT (1.75g/kg, up to maximum of 75g glucose administered).
Change in liver enzymes (ALT, AST, GGT, or ALP) | Six months
  Liver enzymes will be measured using Abbott ARCHITECT Systems
Change in body fat percentage | Six months
  Body fat will be measured using a DXA scanner, by research team members previously trained in DXA measurement.
Change in weight | Six months
  Weight will be measured using an electronic platform scale.
Change in height | Six months
  Height will be measured using a wall mounted stadiometer.
Change in BMI | Six months
  BMI will be calculated mathematically from other outcomes such as height and weight.

OTHER OUTCOMES:
Changes in molecular profiling of gut microbiome | Six months
  Profiling of the gut microbiome will be measured from collected stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Pai, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No